CLINICAL TRIAL: NCT00153738
Title: Effectiveness of Phytosterol Supplementation on Select Indices of Cardiovascular Risk
Brief Title: Phytosterol Supplementation and Cardiovascular Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cooper Institute (Other)
Collaborators: Cargill (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: CI0129
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Hypercholesteremia
Keywords: LDL-C, phytosterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — Phytosterols

INTERVENTIONS:
Drug: phytosterol

SUMMARY:
This study examined the effects of 2.6 g/d of phytosterol ingestion on LDL cholesterol metabolism. It is expected that this dose will significantly reduce LDL cholesterol after 12 weeks of supplementation.

DETAILED DESCRIPTION:
This study examined the effects of 2.6 g/d of phytosterol ingestion on LDL cholesterol metabolism. It is expected that this dose will significantly reduce LDL cholesterol after 12 weeks of supplementation.

The study recruited 72 men and women 20-70 years of age with mild hypercholesteremia (>130 mg/dl LDL-C). They were assigned to 1 of 2 groups. Participants ingested the supplement or a placebo for 12 weeks, with an interim assessment at 6 weeks. Participants agreed to maintain current diet, medication, and exercise habits and to not donate blood during the trial.

ELIGIBILITY:
Inclusion Criteria:

* mild hypercholesteremia, sign informed consent, not donate blood, maintain diet and exercise habits

Exclusion Criteria:

* BMI <18.5 or >34.9, recent blood donation, serious or life-threatening disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72
Dates: Start 2004-03; Study Completion 2005-08

PRIMARY OUTCOMES:
Ingestion of the supplement will result in reduced LDL cholesterol.

CONTACTS AND LOCATIONS:
Overall Officials: Conrad Earnest, PhD, Principal Investigator — The Cooper Institute
Locations (1):
- The Cooper Institute, Dallas, Texas, United States